CLINICAL TRIAL: NCT04438655
Title: Prospective Randomized Clinical Trial on Oral and Intravenous Antibiotic Prophylaxis in Colorectal Surgery (COLORAL1).
Brief Title: Prospective Randomized Clinical Trial on Oral and Intravenous Antibiotic Prophylaxis in Colorectal Surgery.
Acronym: COLORAL1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Alberto Arezzo, Prof., University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Università di TORINO
Record Dates: First submitted 2020-04-18; First posted 2020-06-19 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Surgery
MeSH Terms: interventions — Anti-Infective Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral + Parenteral prophylaxis (Experimental): Oral antibiotic drugs:
  - Bimixin (Neomicin + Bacitracin tablet) 25000 UI + 2500 UI: h. 8-16-24 the day before surgery if the procedure takes place in the morning; h. 16-24-8 if the procedure takes place in the afternoon.
  Systemic antibiotic drugs:
  * Amoxicillin - Clavulanic Acid 2000/200 mg at induction of anesthesia, redosing with prolonged surgery.
  * in case of allergy to penicillin: Clindamycin 600 mg + Gentamycin 2 mg/kg.
  Interventions: Drug: Oral antibiotic drugs; Drug: Parenteral prophylaxis
- Only parenteral prophylaxis (Sham Comparator): * Amoxicillin - Clavulanic Acid 2000/200 mg at induction of anesthesia, redosing with prolonged surgery.
  * in case of allergy to penicillin: Clindamycin 600 mg + Gentamycin 2 mg/kg.
  Interventions: Drug: Parenteral prophylaxis

INTERVENTIONS:
Drug: Oral antibiotic drugs — Oral antibiotic drugs:
  - Bimixin (Neomicin + Bacitracin tablet) 25000 UI + 2500 UI: h. 8-16-24 the day before surgery if the procedure takes place in the morning; h. 16-24-8 if the procedure takes place in the afternoon.
  Arms: Oral + Parenteral prophylaxis
Drug: Parenteral prophylaxis — Amoxicillin - Clavulanic Acid 2000/200 mg at induction of anesthesia, redosing with prolonged surgery.
  in case of allergy to penicillin: Clindamycin 600 mg + Gentamycin 2 mg/kg.

SUMMARY:
Elective colon surgery is considered a clean-contaminated procedure, with a Surgical Site Infection (SSI) rate not inferior to 10%. For many years the role of Mechanical Bowel Preparation (MBP) has been universally recognized as an effective measure to reduce colonic bacterial load and consequently SSI rate, mostly in European Countries. However, in the early 1970s has been demonstrated a further SSI risk reduction in colon surgery if oral non-absorbable antibiotics were added to MBP and for the next 30 years this became the standard of care prior to elective colon surgery, especially in the US. Nowadays, Meta-analyses have demonstrated that MBP does not impact upon postoperative morbidity or mortality, and as such it should not be prescribed routinely. Conversely, recent evidence has suggested that there may be a role for combined MBP and oral antibiotics, or oral antibiotics alone in the prevention of surgical site infection (SSI).

The aim of this trial is to evaluate the efficacy of preoperative oral antibiotics prophylaxis for preventing surgical site infections in elective colorectal surgery.

DETAILED DESCRIPTION:
This study is a Multicenter, Prospective, Randomized, Controlled Trial on preoperative oral antibiotics prophylaxis in colorectal surgery.

INCLUSION & EXCLUSION CRITERIA:

All consecutive patients undergoing elective colorectal resection should be included in the trial.

Exclusion criteria:

* Emergency procedures
* Appendicectomy (unless procedure involves a right hemicolectomy)
* Primarily urological/gynecological or vascular procedure - e.g. ileal conduit, Hartmann's during ovarian surgery, resection during abdominal aortic aneurysm repair.
* Diagnostic laparotomy/laparoscopy without intestinal resection.
* Surgery involving multi-visceral surgery - e.g. pelvic exenteratio
* Controindication for mechanical preparation
* Allergy to used drugs
* Patients who refuse to participate in the study
* Patients with intra-abdominal sepsis before surgery (abscess).
* Patients who received antibiotics for any reason within two weeks prior to surgery.
* Patients who do not comply strictly with the assigned prophylaxis regimen.
* Patients who cannot be followed at least 4 weeks after surgery.

Patients recruitment:

Consecutive eligible patients will be recruited at the outpatient clinic in the participating center by the involved physician (surgeon). All patients fulfilling the inclusion criteria will be informed about the study by the physician. After consent is given, central data acquisition will take place web-based and patients will be randomized in 2 groups and treated according to the study protocol. Patients unable or refusing to provide informed consent will be treated according to current clinical practice.

Primary Outcome:

- Incidence of surgical site infections (superficial or deep)

Secondary Outcomes:

* Perioperative complication
* Anastomotic dehiscence
* Post-operative ileus
* Extra-abdominal complications
* Readmission
* Reoperation
* Length of hospital stay
* Mortality
* Adverse effects of antibiotics (diarrhea, C. difficile infection)

Covariates:

In addition to demographic, procedure and outcome data, the following data will be collected as confounding variables to permit accurate risk adjustment of outcomes.

* The American Society of Anesthesiologists (ASA) score
* Cardiovascular and metabolic co-morbidities (includes chronic obstructive pulmonary disease (COPD), chronic kidney disease (CKD), peripheral vascular disease (PVD) and diabetes mellitus)
* History of previous abdominal surgery
* Preoperative administration of immunosuppressive/steroid therapy
* Preoperative Chemo-RadioTherapy
* Preoperative Albumin Serum Level (g/dL)

Follow-up:

* Patients will be followed for 30 days after surgery. All secondary outcome measures will be recorded if they occurred at any point from post-operative day 0 (day of surgery) to Day 30.
* No change to normal follow-up should take place.
* The follow-up of patients includes a clinical evaluation 30 days after surgical intervention supported by blood analysis (WBC count and CRP), to completely exclude the presence of any infectious complication. Presence of fever and/or WBC count/CRP elevation will require further investigation with radiological imaging and will be considered an infectious post operative complication (SSI or not).

PROJECT TIMELINE:

Data collection will take place in two years. Follow-up data will also be collected for up to 30 days after surgery.

Data Collection and Governance:

Data will be collected and stored online. Communication between the clients and the Server where is hosted the online platform is secured under TLS protocol with an encryption certificate SHA256 with RSA 2048 bits (e 65537). In order to maximize the data protection, the physical HD where is sored the database is encrypted too. Access to the online platform will be possible only previous Login. Each device logged in will be identified and the user will be able to ban the access from a specific device. Each physician will be able to see and modify only the data of patients added from his center. The online platform will check the validity and the correct format of the fields and will generate an excel table to import to the statistic software.

Intervention strategies:

Patients will be randomized to intravenous antibiotic prophylaxis alone or oral antibiotics prepara-tion in association with intravenous antibiotic prophylaxis.

In the group of patients not treated with oral antibiotics standard intravenous prophylaxis will be administered at the time of induction of anesthesia, redosing with prolonged surgery: amoxicil-lin/clavulanic acid 2000/200 mg or, in the event of allergy to penicillin, clindamycin 600 mg + gen-tamycin 2 mg/kg. In case of Chronic Renal Failure dose adjustment will be necessary in presence of Creatinine Clearance respectively <30 ml/min and <60 ml/min in accordance to pharmacologic recommendations.

In the other group oral prophylaxis consists of Bimixin (Neomicin + Bacitracin tablet) 25000 UI + 2500 UI). In the postoperative period no more doses will be administered because the drug is not absorbed by gastrointestinal mucosa and its progression from the stomach to the colon is slowed down by post-operative ileus. In this group of patient standard intravenous antibiotic prophylaxis will be administered at induction of anesthesia.

Any mechanical bowel preparation will be administered, as indicated by each center. Surgeon, anesthesiologist and nurse will know if patient had assumed oral antibiotics and intrave-nous antibiotics or intravenous prophylaxis alone. Data concerning SSI rate, infectious complica-tion other than SSI and not infectious complications will be collected during hospital stay. 30 days after the operation blood tests (WBC, CRP) and clinical evaluation will confirm the absence of any infectious complication.

ELIGIBILITY:
Inclusion criteria:

* Summary: All consecutive patients undergoing colorectal resection should be included.
* Age: Age 18 years or above.
* The general health condition of the patient permits general anesthesia (ASA- classification I-III).
* Absence of allergy to the oral antibiotics employed
* Timing: Elective procedures.
* Technique: Open, laparoscopic, laparoscopic-assisted or laparoscopic converted to open.
* Returns to theatre: Each patient should only be included in the study once. Return to theatre during the same admission or follow up should be collected as a complication.
* Included procedures: Any colorectal resection (See Appendix B).
* Mechanical Bowel Preparation: Any mechanical bowel preparation (as indicated by each centre).

Exclusion criteria:

* Emergency procedures
* Appendicectomy (unless procedure involves a right hemicolectomy)
* Primarily urological/gynecological or vascular procedure - e.g. ileal conduit, Hartmann's during ovarian surgery, resection during abdominal aortic aneurysm repair.
* Diagnostic laparotomy/laparoscopy without intestinal resection.
* Surgery involving multi-visceral surgery - e.g. pelvic exenteratio
* Controindication for mechanical preparation
* Allergy to used drugs (neomycin sulfate, amoxicillin-clavulanic acid)
* Patients who refuse to participate in the study
* Patients with intra-abdominal sepsis before surgery (abscess).
* Patients who received antibiotics for any reason within two weeks prior to surgery.
* Patients who do not comply strictly with the assigned prophylaxis regimen.
* Patients who cannot be followed at least 4 weeks after surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Wound infection | up to 30 days after surgery
  Incidence of surgical site infections (superficial or deep)

SECONDARY OUTCOMES:
Perioperative complication | up to 30 days after surgery
  Incidence of any preoperative complication, assessed as clinically detected
Anastomotic dehiscence | up to 30 days after surgery
  Incidence of anastomotic dehiscence, assessed as clinically detected
Post-operative ileus | up to 30 days after surgery
  length of post-operative ileus, assessed as time to first flatus
Extra-abdominal complications | up to 30 days after surgery
  Iatrogenic problems, bleeding, Cardiac- nephrological - respiratory and gastrointestinal complications
Readmission | up to 30 days after surgery
  incidence of readmission to hospital ward
Reoperation | up to 30 days after surgery
  incidence of reoperation
Length of hospital stay | up to 30 days after surgery
  Hospital stay since colorectal surgery
Mortality | up to 30 days after surgery
  incidence of death for any cause
Adverse Drug Reactions | up to 30 days after surgery
  Allergic reactions / Intolerance

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Arezzo, Prof., Principal Investigator — University of Turin, Italy
Locations (1):
- Università degli studi di Torino, Turin, Torino, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American College of Surgeons. National Surgical Quality Improvement Program Semi-annual report. 2009. Available at: https://acsnsqip.org/login/default.aspx.
- [Background] Arriaga AF, Lancaster RT, Berry WR, Regenbogen SE, Lipsitz SR, Kaafarani HM, Elbardissi AW, Desai P, Ferzoco SJ, Bleday R, Breen E, Kastrinakis WV, Rubin MS, Gawande AA. The better colectomy project: association of evidence-based best-practice adherence rates to outcomes in colorectal surgery. Ann Surg. 2009 Oct;250(4):507-13. doi: 10.1097/SLA.0b013e3181b672bc. PMID 19734778
- [Background] Csikesz NG, Nguyen LN, Tseng JF, Shah SA. Nationwide volume and mortality after elective surgery in cirrhotic patients. J Am Coll Surg. 2009 Jan;208(1):96-103. doi: 10.1016/j.jamcollsurg.2008.09.006. Epub 2008 Oct 31. PMID 19228510
- [Background] Finlayson EV, Goodney PP, Birkmeyer JD. Hospital volume and operative mortality in cancer surgery: a national study. Arch Surg. 2003 Jul;138(7):721-5; discussion 726. doi: 10.1001/archsurg.138.7.721. PMID 12860752
- [Background] Nichols RL, Broido P, Condon RE, Gorbach SL, Nyhus LM. Effect of preoperative neomycin-erythromycin intestinal preparation on the incidence of infectious complications following colon surgery. Ann Surg. 1973 Oct;178(4):453-62. doi: 10.1097/00000658-197310000-00008. No abstract available. PMID 4743867
- [Background] Slim K, Vicaut E, Launay-Savary MV, Contant C, Chipponi J. Updated systematic review and meta-analysis of randomized clinical trials on the role of mechanical bowel preparation before colorectal surgery. Ann Surg. 2009 Feb;249(2):203-9. doi: 10.1097/SLA.0b013e318193425a. PMID 19212171